CLINICAL TRIAL: NCT06471907
Title: Comparison of Pain Relief and Peripheral Perfusion Index Using Different Volume of Erector Spinae Plane Block
Brief Title: Comparison of Pain Relief and Peripheral Perfusion Index
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-04-007-003
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Erector Spinea Plane Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 ml lumbar ESPB group (Placebo Comparator): lumbar ESPB was performed with 10 ml of local anesthetics
  Interventions: Procedure: erector spinae plane block
- 20 ml lumbar ESPB group (Experimental): lumbar ESPB was performed with 20 ml of local anesthetics
  Interventions: Procedure: erector spinae plane block

INTERVENTIONS:
Procedure: erector spinae plane block — fascial plane injection using ultrasound

SUMMARY:
The primary endpoint of this study is to compare the pain relief and peripheral perfusion index using different volume of local anesthetics in erector spinae plane block.

DETAILED DESCRIPTION:
The erector spinae plane block (ESPB) is a less invasive, safer, and technically easy alternative procedure to conventional neuraxial anesthetic techniques. In contrast to common neuraxial techniques such as paravertebral and epidural injections, the ESPB targets an interfascial plane which is far from the spinal cord, root, and pleura. First applied to thoracic neuropathic pain, currently ESPB is being applied to postoperative pain control and includes variable clinical situations. In the abdomen and thoracic wall, thoracic ESPB can be applied for pain control after cardiac surgery, video-assisted thoracic surgery, laparoscopic cholecystectomy, and thoracotomy. Recently, favorable postoperative pain control after lumbar spinal or lower limb surgeries has been reported with lumbar ESPB. In addition, ESPB has also been used for chronic pain conditions in the upper and lower extremities. To investigate the possible mechanism of action of the ESPB, many previous studies have focused on examining the physical spread of the injected agent. Commonly, contrast dye injections in human cadavers have been utilized to assess the spread level. Physical spread level was determined using various methods including direct dissection or sectioning, computed tomography (CT), thoracoscopic inspection, or magnetic resonance imaging (MRI) with radiocontrast injection. Apart from human cadaver studies, physical spread level has been evaluated in alive patients using a variable volume of local anesthetics mixed with radiocontrast. Perfusion index is an indirect method which can present the degree of peripheral perfusion. Moreover, it is known as a more sensitive measurement tool than the rise of skin temperature. The apply of perfusion index is very simple and noninvasive. The degree of PI increase has been used to determine the success of peripheral nerve block. The volume of local anesthetics has been used 10-30 ml. However, most effective dosage with proper pain relief has never been suggested.

ELIGIBILITY:
Inclusion Criteria:

* lumbar disc herniation
* lumbar foraminal stenosis
* lumbar central stenosis
* lumbar spondylolisthesis
* numerical rating scale > 4
* back pain functional scale < 45
* duration of pain > 1 mon
* patients who can fully understand all items described in back pain functional scale

Exclusion Criteria:

* Allergy to local anesthetics or contrast medium
* Pregnancy
* Spine deformity
* Prior history of lumbar spine surgery
* No previous lumbar MRI or CT
* Patients with coagulation abnormality

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale changes among 5 times period | Baseline, 2 weeks, 4 weeks, 8 weeks after the completion of erector spine plane block
  minimum (1) and maximum value (10), lower score means better outcome

SECONDARY OUTCOMES:
back pain functional scale among 3 times period | Baseline, 4 weeks, 8 weeks after the completion of erector spine plane block
  minimum (0) and maximum value (60), higher score means better outcome
Perfusion index changes among 4 times period | baseline, 10minutes after ESPB, 20 minutes after ESPB, 30 minutes after ESPB
  erfusion index changes after lumbar ESPB among 4 times period

CONTACTS AND LOCATIONS:
Locations (1):
- Hong ji HEE, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No